CLINICAL TRIAL: NCT01153230
Title: Study of Frequencies of Histo-pathological Findings in Paraquat Poisoned Patients
Brief Title: Frequencies of Histo-pathological Findings in Patients With Paraquat Toxicity
Status: Completed | Type: Observational
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Other Study IDs: ASD-1213-4
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2008-11

CONDITIONS: Paraquat Toxicity
Keywords: PQ

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- poisoned patient: after patients died the pathological findings evaluated with autopsy

SUMMARY:
The purpose of this study is to determine frequencies of histo-pathological findings in dead poisoned patients and evaluate their relationships with age, gender, dosage of poisoning, time of admission and time of death.

DETAILED DESCRIPTION:
Acute poisoning of paraquat which is taken either to commit suicide or by mistake has become a social problem in world. The present study was conducted to determine frequencies of histo-pathological findings in dead poisoned patients and evaluate their relationships with age, gender, dosage of poisoning, time of admission and time of death.

ELIGIBILITY:
Inclusion Criteria:

* every patients who dithionate test were positive

Exclusion Criteria:

* nothing

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: forty two poisoned patients
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2002-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
histo-pathological findings | 1 day after patient died
  for evaluate of this outcome we gather autopsy data

SECONDARY OUTCOMES:
age | 5 min after admission time
  we gathered demogeraphic data such as age
gender | 5 min after admission time
  we gathered demographic data such as gender
dosage of poisoning | 5 min after admission time
  we gathered historical data then estimated dosage of paraquat ingestion

CONTACTS AND LOCATIONS:
Overall Officials: hamidreza shemshaki, MD, Study Chair — MD,research comittee
Locations (1):
- Noor university hospital, Isfahan, Iran